CLINICAL TRIAL: NCT00553657
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study to Evaluate the Effect of Standardization of Fluid Intake on the Variability of Measured Voiding Parameters in Female Patients With Idiopathic Overactive Bladder
Brief Title: The Study To Test The Effect of Standardization Of Fluid Intake In Female Patients With Overactive Bladder
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Study Director, GSK
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: BKB105190
Record Dates: First submitted 2007-11-02; First posted 2007-11-05 (Estimated); Last update posted 2010-10-26 (Estimated); Status verified 2010-10

CONDITIONS: Overactive Bladder
Keywords: Experimental Medicine
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Tolterodine Tartrate; Pharmaceutical Preparations

INTERVENTIONS:
Drug: DETROL LA (drug)

SUMMARY:
The purpose of this study is to determine if standardizing fluid intake in a clinic setting will reduce variability of individual voiding parameters and potentially serve as a way to limit patient exposure in the initial assessment of efficacy of compounds being developed for Overactive Bladder.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants will be females who are 18 years of age or older, with Overactive Bladder as evidenced by daily episodes of urgency without incontinence, which may be associated with frequency or nocturia but without bladder pain. At screening, eligible patients must report frequency, defined as at least 8 micturitions per 24 hour period.
* Eligible patients must have signed the informed consent and must meet all inclusion and exclusion criteria as determined during the screening visit.

Exclusion Criteria:

* Any abnormality identified on the screening examination or any other medical condition or circumstance making the patient unsuitable for participation in the study based on the Investigator's and Medical Monitor's assessment
* Any contraindication to Detrol LA or other anti-muscarinic medications
* Inability to consume 10 cc/kg of fluid within 30 minutes
* Regular alcohol consumption averaging ³7 drinks/week for women (1 drink = 100mL of wine or 285mL of beer or 30mL of hard liquor)
* Positive urine drug or alcohol at screening at screening
* Average blood pressure measurements systolic ≥140 or diastolic ≥90 at screening at screening
* QTcB value ≥ 450 msec at screening
* Poorly-controlled diabetes mellitus or hypertension, as evidenced by a change in medication within the 2 months prior to initiation of the study
* History of urinary retention or gastric retention
* Known history of narrow-angle glaucoma
* History of QT prolongation
* Known reduction in hepatic or renal function
* Concomitant Use of loop diuretics (eg. Furosemide)
* Concomitant use of a medication that is a potent inhibitor of CYP3A4
* Class IA or Class III antiarrhythmic medications
* Patient is unable and/or unwilling to adhere to Lifestyle Guidelines
* For women of child bearing potential, a positive serum β-hCG at screening or pre-dose, or an unwillingness to agree to adequate contraception from the time of screening until the completion of the study:
* Positive for hepatitis C antibody, hepatitis B surface antigen or HIV at screening.
* Presence of urinary tract infection within 4 weeks of screening.
* Post-void residual of >150 mL (bladder ultrasound).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2007-08; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Variability of change from baseline in mean volume per void measured on 3 consecutive days. | 3 consecutive days

SECONDARY OUTCOMES:
Mean change from baseline in volume voided per void. Percent and actual change from baseline in maximum volume voided, number of micturitions, number of incontinence episodes, number of urgency episodes, and time to first void on 3 consecutive days. | 3 consecutive days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Randwick, Sydney, New South Wales, Australia

REFERENCES:
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401